CLINICAL TRIAL: NCT07163598
Title: Peripheral Nerve Block Anesthesia Improves Older Patients' Postoperative Early Recovery Outcomes After Total Hip Arthroplasty: a Retrospective Clinical Trial
Brief Title: PNB Anesthesia Improves Older Patients' Postoperative Early Recovery Outcomes After Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Professor, RenJi Hospital
Other Study IDs: KY2022-066-B
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Arthroplasty (THA); Femoral Neck Fractures
Keywords: Total hip arthroplasty; peripheral nerve block anesthesia; QoR-40 score
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- peripheral nerve block group
  Interventions: Other: No Intervention: Observational Cohort
- general anesthesia group
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This study is a observational cohort study, and we have no intervention.

SUMMARY:
Early postoperative rehabilitation is an important issue for total hip arthroplasty, especially in older patients. This retrospective clinical trial is to assess the impact of peripheral nerve block anesthesia versus general anesthesia in older patients' early recovery outcomes after total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged over 60 years; 2. patients underwent total hip replacement; 3. the surgery was done with ultrasound-guided nerve block alone or under general anesthesia.

Exclusion Criteria:

1. patients who failed to the nerve block and were changed to general anesthesia for the operation; 2. patients who lost contact 3 months after surgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older patients who visited Renji Hospital affiliated with Shanghai Jiao Tong University school of medicine for total hip arthroplasty were enrolled between 11/2020 and 12/2024.
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
postoperative QoR-40 scores | 1-day and 3-month

CONTACTS AND LOCATIONS:
Locations (1):
- RenjiH, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No